CLINICAL TRIAL: NCT04213976
Title: Ostomy in Continuity or Conventional Ileostomy for Complex Pediatric Intestinal Diseases: a Retrospective Multicentric Analysis
Brief Title: Ostomy in Continuity or Conventional Ileostomy: a Retrospective Multicentric Analysis
Acronym: StomaPed
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019/10
Record Dates: First submitted 2019-12-19; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Intestinal Obstruction; Gastroschisis; Enterocolitis, Necrotizing; Hirschsprung Disease
Keywords: ileostomy; enteral nutrition; complications of stoma
MeSH Terms: conditions — Intestinal Obstruction; Gastroschisis; Enterocolitis, Necrotizing; Hirschsprung Disease | interventions — Ileostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ileostomy in continuity: Paediatric patients having had an ileostomy in continuity as part of the treatment for a complex intestinal obstruction, as described by Santulli or by Bishop-Koop.
  Interventions: Procedure: Ileostomy
- Conventional ileostomy: Paediatric patients having had a loop ileostomy as part of the treatment for a complex intestinal obstruction.
  Interventions: Procedure: Ileostomy

INTERVENTIONS:
Procedure: Ileostomy — Use of an ileostomy to decompress the proximal bowel, perfored either as a conventional loop ileostomy or as described by Santulli et al. or by Bishop and Koop.
  Other Names: Loop ileostomy; Santulli ileostomy; Bishop-Koop ileostomy

SUMMARY:
Surgical procedures for complex intestinal neonatal and paediatric diseases may require the use of an ostomy, in order to discharge the upper intestine. The traditional loop ileostomy has recently be challenged by ileostomies in continuity, either the Santulli or the Bishop-Koop one, that both decompresses the proximal dilated bowel and allow intestine fluid to pass through the underlying ileal anastomosis. Nevertheless, to date, no evaluation of their indications, complications and potential benefits has been made.

The aim of this study is to retrospectively compare the outcomes of loop ileostomies and ileostomies in continuity in a paediatric population.

It is thus expected to better define the specific indications for these different types of ileostomies in the paediatric and neonatal population.

DETAILED DESCRIPTION:
The methodology used will be a retrospective non interventional study of the cohorts of paediatric patients having had one or more ileostomies performed in one of the surgical centers participating in this study, between 2007, january the 1st and 2019, august the 31th.

The main outcome will be the duration (days) between full refunctionalization of the bowel in the groups of conventional ileostomy or ostomy in continuity, as assessed by the end of parenteral nutrition or the closure of the stoma.

Secondary outcomes will include (1) the number and type of complications directly related to the stoma and/or to intestinal complications; (2) the comparison of the results obtained by Santulli and Bishop-Koop ileostomies; (3) a sub-group analysis of the outcomes in the different underlying pathologies.

ELIGIBILITY:
Inclusion Criteria:

* all patient aged 16 or less having had one or more ileostomy created as part of its care for an intestinal obstruction, between 2007/01/01 and 2019/08/31. If a patient requires more than one ileostomy, each new stoma will be analysed as a new entry in the study.
* patients having been operated in one of the paediatric surgical department participating in this study.

Exclusion Criteria:

* refusal or absence on consent of the patient and/or their legal representative to participate to the study.
* patient who had an ileostomy created in another center than the ones participating in the present study.

Ages: 1 Minute to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns and children presenting with complex intestinal obstruction and requiring the use of an ileostomy to discharge the upper intestine as part of surgical care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Delay before full refunctionalization of the small intestine | through study completion, an average of 6 months
  Mean delay before full enteral nutrition after the creation of the ileostomy, as assessed by either the end of the use of parenteral nutrition, or by closure of the ileostomy.

SECONDARY OUTCOMES:
Clinical description of the sub-groups of patients with ostomy in continuity | through study completion, an average of 6 months
  Clinical description of the patients (underlying disease, demographics, nutritional outcomes, medical and surgical complications) having had a Santulli or a Bishop-Koop ostomy.
Comparative analysis of the complications of ostomies | through study completion, an average of 6 months
  Number and type of complications encountered after loop ileostomy and after ostomy in continuity
Subgroup analysis of the patients according to their underlying pathology | through study completion, an average of 6 months
  Comparative analysis of the efficacy and complication rates of the different types of stoma in subgroups of patients, according to their underlying pathology

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Schmitt, MD, PhD, Principal Investigator — University Hospital of Angers
Locations (5):
- France (5):
  - University Hospital of Brest, Brest
  - University Hospital of Nantes, Nantes
  - Necker Enfants Malades Hospital, Paris
  - University Hospital of Rennes, Rennes
  - University Hospital of Tours, Tours

REFERENCES:
- [Result] BISHOP HC, KOOP CE. Management of meconium ileus; resection, Roux-en-Y anastomosis and ileostomy irrigation with pancreatic enzymes. Ann Surg. 1957 Mar;145(3):410-4. doi: 10.1097/00000658-195703000-00017. No abstract available. PMID 13403593
- [Result] SANTULLI TV, BLANC WA. Congenital atresia of the intestine: pathogenesis and treatment. Ann Surg. 1961 Dec;154(6):939-48. No abstract available. PMID 14497096
- [Result] Sehgal S, Sandler AD, Alfred Chahine A, Mohan P, Torres C. Ostomy in continuity: A novel approach for the management of children with complex short bowel syndrome. J Pediatr Surg. 2018 Oct;53(10):1989-1995. doi: 10.1016/j.jpedsurg.2018.02.059. Epub 2018 Mar 4. PMID 29602547